CLINICAL TRIAL: NCT00003192
Title: A Phase II Trial of 9-Aminocamptothecin (NSC 603071) Administered as a 120-Hour Continuous Infusion in Patients With Previously Untreated Gastric Cancer
Brief Title: Aminocamptothecin in Treating Patients With Stomach Cancer or Cancer of the Esophagus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9025; UCCRC-9025; NCI-T97-0013
Record Dates: First submitted 1999-11-01; First posted 2004-03-30 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; adenocarcinoma of the stomach
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm A (Experimental): 9-aminocamptothecin (25 mcg/m2/hr x 120hrs, days 1-5 and 8-12 of each 3 week cycle)
  Interventions: Drug: aminocamptothecin

INTERVENTIONS:
Drug: aminocamptothecin
  Other Names: 9-AC

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of aminocamptothecin in treating patients with locally advanced, metastatic, or recurrent cancer of the stomach or esophagus.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the objective response rate of a 120 hour continuous infusion of aminocamptothecin (9-AC) in chemotherapy naive patients with adenocarcinoma of the stomach or gastroesophageal junction. II. Characterize the nature of the toxicity of 9-AC on this schedule in this patient population. III. Determine the duration of response, time to progression, and survival of this patient population. IV. Study the pharmacokinetics and pharmacodynamics of 9-AC on this schedule in these patients.

OUTLINE: This is an open label, multicenter study. Patients receive intravenous aminocamptothecin by continuous infusion over 120 hours on days 1-5 and 8-12 followed by 1 week of rest for a 3 week cycle. Therapy continues for a minimum of 6 weeks (2 full cycles) unless there are unacceptable toxic effects or rapid disease progression. Dose escalation may occur in patients who complete 3 cycles of therapy without unacceptable toxicity. All patients will be followed for survival.

PROJECTED ACCRUAL: This study will accrue 14-40 patients within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed, locally advanced, metastatic or recurrent adenocarcinoma of the stomach or gastroesophageal junction Measurable disease CNS metastases allowed provided that patient has other sites of measurable disease, is neurologically stable, and is receiving no concurrent anticonvulsant therapy

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: CALGB 0-2 Life expectancy: Not specified Hematopoietic: WBC at least 3500/mm3 Absolute neutrophil count at least 1500/mm3 Platelet count at least 100,000/mm3 (no platelet transfusion within 7 days) Hemoglobin at least 9 g/dL Hepatic: Total bilirubin no greater than 1.5 mg/dL Transaminases no greater than 2.5 times upper limit of normal (ULN) (no greater than 5 times ULN if liver metastases) Renal: Creatinine no greater than 1.5 mg/dL OR Creatinine clearance at least 60 mL/min Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No concurrent uncontrolled medical or psychiatric condition No active uncontrolled infection No prior malignant disease within the past 5 years except curatively treated non-melanoma skin cancer and carcinoma in situ of the cervix

PRIOR CONCURRENT THERAPY: Biologic therapy: No concurrent prophylactic growth factors Chemotherapy: One prior adjuvant or neoadjuvant 5-FU-based chemotherapy regimen allowed At least 4 weeks since prior adjuvant or neoadjuvant chemotherapy (6 weeks if nitrosoureas or mitomycin) and recovered No prior therapy with a topoisomerase I inhibitor No other concurrent chemotherapy Endocrine therapy: Not specified Radiotherapy: One prior radiotherapy regimen allowed No prior radiation therapy to only site of measurable disease At least 4 weeks since prior radiation therapy and recovered No concurrent palliative radiation therapy Surgery: Not specified Other: See Disease Characteristics No other concurrent investigational antineoplastic therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 1998-03; Primary Completion 2002-02 (Actual); Study Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Objective response rate Objective response rate Objective response rate Objective response rate | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Hedy L. Kindler, MD, Study Chair — University of Chicago
Locations (7):
- United States (7):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, S.C., Decatur, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Central Illinois Hematology Oncology Center, Springfield, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Michiana Hematology/Oncology P.C., South Bend, Indiana